CLINICAL TRIAL: NCT00601952
Title: Information Processing Modification in PTSD
Brief Title: Information Processing Modification in PTSD (Oct. 18)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, Nader Amir, Professor, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PT074970; PT074970 (Other: Department of Defense)
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Results first posted 2014-02-04 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2009-07

CONDITIONS: Stress Disorders, Post-traumatic
Keywords: post traumatic stress disorder; cognitive bias; attention; combat
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Attention Bias Modification (ABM) (Experimental): The ABM comprised a probe detection paradigm described above, modified to facilitate the allocation of attention away from threatening material. In this task, the probe always replaced the neutral word. Stimuli comprised a different set of 12 threat-neutral word pairs different than those used in the attention bias assessment. Participants completed 288 training trials: 2 (probe type) x 2 (probe location) x 2 (threat location) x 12 (threat-neutral word pairs) x 3 (repetition). Thus, although there were no explicit instructions to direct attention away from threat words, on all trials, the position of the neutral word indicated the position of the probe.
  Interventions: Behavioral: Attention Bias Modification (ABM)
- 2 Attention Control Condition (ACC) (Placebo Comparator): The ACC condition was identical to the ABM procedure with the exception that the probe appeared with equal frequency in the position of the threat and neutral words, such that attention was neither trained towards nor away from threat.
  Interventions: Behavioral: Attention Control Condition (ACC)

INTERVENTIONS:
Behavioral: Attention Bias Modification (ABM) — The ABM comprised a probe detection paradigm described above, modified to facilitate the allocation of attention away from threatening material. In this task, the probe always replaced the neutral word. Stimuli comprised a different set of 12 threat-neutral word pairs different than those used in the attention bias assessment. Participants completed 288 training trials: 2 (probe type) x 2 (probe location) x 2 (threat location) x 12 (threat-neutral word pairs) x 3 (repetition). Thus, although there were no explicit instructions to direct attention away from threat words, on all trials, the position of the neutral word indicated the position of the probe.
  Arms: 1 Attention Bias Modification (ABM)
Behavioral: Attention Control Condition (ACC) — The ACC condition was identical to the ABM procedure with the exception that the probe appeared with equal frequency in the position of the threat and neutral words, such that attention was neither trained towards nor away from threat.
  Arms: 2 Attention Control Condition (ACC)

SUMMARY:
The purpose of this study is to determine whether a computerized intervention designed to change the nature of attention biases will be effective in reducing the symptoms of post traumatic stress disorder (PTSD) in American combat veterans returning from the wars in Afghanistan and Iraq.

DETAILED DESCRIPTION:
Operation Iraqi Freedom (OIF) and Operation Enduring Freedom (OEF) in Afghanistan are the largest sustained ground operations since the Vietnam War, and the psychological effects of combat on military personnel can be devastating. Approximately thirty percent of returning veterans present with mental health problems. Posttraumatic stress disorder (PTSD) is the most common problem in this group (52% of overall diagnoses). This translates into PTSD prevalence rates of 12% in Afghani veterans and 19% for Iraqi veterans, rates that are two to three times higher than the overall lifetime prevalence rate in the general population (8%). Of those veterans screened positive for mental health problems 70% have not received any mental health services. Therefore, even for individuals identified as having psychological problems the majority are not receiving any help. Prevention and treatment of this disorder represents one of the greatest challenges facing government officials and health care professionals working with combat veteran populations.

PTSD often manifests after the experience of a trauma in which individuals undergo threat of injury or death to themselves or others. The experience includes intense feelings of fear, helplessness, and/or horror. Symptoms of this disorder are often chronic lasting for years. Those with PTSD are likely to experience problems across several life domains including higher rates of divorce, problems raising children, and engaging in domestic violence. They are also more likely to suffer from other mental health problems including depression, substance abuse, and generalized anxiety disorder. Moreover, they tend to report less life satisfaction, experience poorer physical health, earn less money, and change jobs frequently.

Although effective treatments do exist for PTSD, as many as 44% of individuals do not respond to psychosocial and pharmacological treatments. Thus, there is a clear need to develop highly effective and efficient treatments for PTSD. Researchers have established a relationship between PTSD and difficulty disengaging attention from threat relevant inforamtion. This knowledge; however, has not been translated into more effective treatments for this disorder. This three-year proposal aims to test a computerized treatment for PTSD in a double-blind, placebo-controlled study that would bridge research on attention bias and treatment development. Those in the active condition will receive a computer-delivered attention modification program (AMP) designed to enhance attention disengagement from threatening stimuli. The AMP protocol includes six weeks of biweekly sessions in which participants see 240 trials consisting of the various combinations of probe type (E or F), probe position (top or bottom), and word type (Neutral or Trauma). Of the 240 trials, 48 include only neutral words: 2 (probe type) X 2 (probe position) X 12 (word pairs). The remaining 192 trials include one neutral word and one trauma word: 2 (probe type) X 2 (probe position) X 2 (repetitions) X 24 (word pairs). On trials where participants see one neutral word and one trauma word (i.e., 80% of the trials), the probe always follows the neutral word. Thus, although there is no specific instruction to direct attention away from threat word, on 80% of the trials the position of the threat word indicates the position of the probe (i.e., in the location opposite the threat word). The placebo condition (PC) will be identical to the AMP condition except that during the presentation of threat-neutral word pairs, the probe will appear with equal frequency in the position of threat and neutral words. Thus, neither threat nor neutral words have signal value. We have used a very similar training procedure to successfully establish a pattern of enhanced attention disengagement to threat words in our pilot studies.

We present the results from 2 clinical trials demonstrating the efficacy of attention modification programs (AMP) in ameliorating symptoms of anxiety. Specifically, we report results from studies of individuals with generalized social phobia (GSP; n=32) and generalized anxiety disorder (GAD; n=24) demonstrating the effectiveness of the procedures described in this proposal. In brief, our intervention was effective in: a) changing biased attention, b) reducing clinical symptoms of anxiety, c) maintaining its effects in up to one year follow-up. This efficient and efficacious technique for changing attention bias in anxiety can provide a low-cost, easy to administer treatment that is grounded in basic cognitive science that may help reduce suffering in individuals with anxiety. The goal of the current proposal is to extend these findings to the highly related disorder of PTSD, and to examine the generalizability of the results to individuals with comorbid conditions. In the current proposal we will test two hypotheses: 1) Individuals with PTSD completing the AMP will show a larger reduction in their attention bias to threat compared to the placebo group, 2) Individuals with PTSD completing AMP will show a larger reduction in anxiety symptoms compared to the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Primary DSM-IV-TR Axis I diagnosis of post-traumatic stress disorder
* Combat veteran from Iraq and/or Afghanistan

Exclusion Criteria:

* No change in medication type or dose during the twelve weeks prior to treatment
* No current psychotherapy
* No evidence of suicidal intent
* No evidence of current substance dependence in the past 6 months
* No evidence of current or past schizophrenia, bipolar disorder, or organic mental disorder

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nader Amir, PhD, Principal Investigator — San Diego State University
Locations (1):
- Center for Understanding and Treating Anxiety, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 Attention Bias Modification (ABM): The ABM comprised a probe detection paradigm, modified to facilitate the allocation of attention away from threatening material. In this task, the probe always replaced the neutral word. Stimuli comprised a different set of 12 threat-neutral word pairs different than those used in the attention bias assessment. Participants completed 288 training trials: 2 (probe type) x 2 (probe location) x 2 (threat location) x 12 (threat-neutral word pairs) x 3 (repetition). Thus, although there were no explicit instructions to direct attention away from threat words, on all trials, the position of the neutral word indicated the position of the probe.
Period: Overall Study
Arm/Group | 1 Attention Bias Modification (ABM) | 2 Attention Control Condition (ACC)
Started | 14 | 17
Completed | 12 | 17
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Attention Bias Modification (ABM) | 2 Attention Control Condition (ACC) | Total
Number analyzed (Participants) | 14 | 17 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 17 | 31
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 13 | 16 | 29
Region of Enrollment [Number; unit: participants]
  United States | 14 | 17 | 31

OUTCOME MEASURES:

1. Primary Outcome: Post-Traumatic Stress Disorder Checklist-Military Version (PCL-M)
Description: The PCL-M is a 17-item questionnaire that assesses the severity of PTSD symptoms using a 5-point Likert scale ranging from "not at all" to "extremely," with a minimum score of 17 and a maximum score of 85 (Weathers, Litz, Herman, Huska, & Keane, 1993). Participants are asked to rate to what extent they experienced PTSD symptoms over the previous month due to prior combat experiences. The military version of the PCL (PCL-M) refers specifically to a traumatic military related event (Weathers, Litz, Huska, & Keane, 1994). Research suggests that the PCL-M has good test-retest reliability (r = .70) and internal consistency (alpha = .97; Weathers et al., 1993).
Time Frame: Pre, Post, Followup
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 Attention Bias Modification (ABM) | 2 Attention Control Condition (ACC)
Number analyzed (Participants) | 12 | 17
units on a scale
  Pre-Treatment | 57.14 (12.48) | 61.33 (11.09)
  Post-Treatment | 52.21 (18.01) | 53.78 (18.31)

ADVERSE EVENTS:
Arm/Group | 1 Attention Bias Modification (ABM) | 2 Attention Control Condition (ACC)
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/17
Other Adverse Events (participants affected / at risk) | 0/14 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes